CLINICAL TRIAL: NCT05799924
Title: The Study on the Therapeutic Effect and Mechanism of Transcutaneous Acupoint Electrical Stimulation in Female
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Honglan Zhu (Other)
Responsible Party: Sponsor-Investigator, Honglan Zhu, Chief physician，OBGYN, Peking University People's Hospital
Organization: Peking University People's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RDL2022-47
Record Dates: First submitted 2023-02-21; First posted 2023-04-05 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-04

CONDITIONS: Dysmenorrhea
Keywords: Dysmenorrhea; acupuncture; TEAS
MeSH Terms: conditions — Dysmenorrhea

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Women with dysmenorrhea treated with TEAS (Experimental): The transcutaneous electrical acupoint stimulator applied alternating current (including sine wave, pulse wave and modulation wave) with frequency of 2 ~ 100Hz and intensity of 10-20mA to stimulate corresponding acupoints through skin electrodes. The stimulated acupoints include Hegu acupoints, Luogong acupoints, Neiguan acupoints and Waiguan acupoints.
  Interventions: Device: Transcutaneous electrical acupoint stimulation
- Women with dysmenorrhea receiving medication (Active Comparator): Take NSAIDs or birth control pills every six hours during your period when you feel unbearable pain.
  Interventions: Drug: non steroidal anti inflammatory drugs

INTERVENTIONS:
Device: Transcutaneous electrical acupoint stimulation — The transcutaneous electrical acupoint stimulator applied alternating current (including sine wave, pulse wave and modulation wave) with frequency of 2 ~ 100Hz and intensity of 10-20mA to stimulate corresponding acupoints through skin electrodes. The stimulated acupoints include Hegu acupoints, Luogong acupoints, Neiguan acupoints and Waiguan acupoints.
  Arms: Women with dysmenorrhea treated with TEAS
Drug: non steroidal anti inflammatory drugs — Hormonal contraception can suppress ovulation, NSAIDS can ease pain
  Other Names: Short-acting birth control pills
  Arms: Women with dysmenorrhea receiving medication

SUMMARY:
The goal of this clinical trial is to investigate the use of TEAS on female patients with dysmenorrhea. The main questions it aims to answer are:

Questions 1：Effect of TEAS on dysmenorrhea Questions 2：Mechanism of TEAS in treatment of dysmenorrhea Participants will wear TEAS devices to treat dysmenorrhea during menstruation The participants in the control group were treated with oral medication for dysmenorrhea

DETAILED DESCRIPTION:
Dysmenorrhea is a common female disease, with an incidence about 20-40% in female, affecting the living quality of the patients. The treatment of dysmenorrhea usually includes hormone drugs to suppress ovulation, and oral non-steroidal anti-inflammatory drugs to relieve pain, but symptoms would relapse after drugs withdrawal. While long-term use of these drugs may cause endocrine disorders, even affect the normal preparation of pregnancy. Recent studies have shown that dysmenorrhea is related to many factors such as immune and neuroendocrine changes. Transcutaneous electric acupoint stimulation (TEAS) is a new therapeutic method derived from traditional acupuncture therapy. In this method, the electrode placed on the surface of the skin of acupoints is used to guide the stimulating current into the body and stimulate the acupoints to achieve the goal of treatment, and can effectively relieve the pain of patients by replacing the traditional mechanical stimulation of hand-twisting needles. The aim of this study is to treat dysmenorrhea in women with TEAS, and to observe the therapeutic effect of TEAS, at the same time, prostaglandins, pain-related factors and immune-related factors were detected in dysmenorrhea women before and after treatment to study the mechanism.

ELIGIBILITY:
Inclusion Criteria:

1. there are symptoms of dysmenorrhea, the duration is more than or equal to 6 months；
2. regular menstruation, menstrual cycle 21 ~ 35 days, menstrual period 3 ~ 7 days.

Exclusion Criteria:

1. dysmenorrhea caused by abnormality and obstruction of reproductive tract；
2. preparing for pregnancy or being pregnant；
3. endometriosis or adenomyosis with surgical indication；
4. taking NSAIDs within one month or receiving immunosuppressive therapy within three months；
5. implantation of pacemaker or other implanted medical electronic devices；
6. high frequency surgical equipment, artificial heart and lung, medical shortwave and microwave therapeutic apparatus were used；
7. scarring or skin damage at the site of irritation；
8. refused to sign the informed consent form.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 240 (Estimated)
Dates: Start 2023-02-21 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale | six months
  The self-rating scale was used to describe the changes of dysmenorrhea symptoms before and after the intervention, with a total score of 0-10, and the greater the number, the more severe the pain.
the Cox Menstrual Symptom Scale | six months
  The self-rating scale was used to describe the changes of dysmenorrhea symptoms before and after the intervention, with the total score ranging from 0 to 100. The greater the number, the more severe the pain.
Work Productivity and Activity Impairment | six months
  The self-rating scale was used to describe the changes of dysmenorrhea symptoms before and after the intervention, with the total score ranging from 0 to 100. The greater the number, the more severe the pain.
Hamilton Anxiety Scale | six months
  The self-rating scale was used to describe the changes of dysmenorrhea symptoms before and after the intervention, with the total score ranging from 0 to 100. The greater the number, the more severe the pain.

SECONDARY OUTCOMES:
Changes in prostaglandins secretion level | six months
  PGF2α is a marker molecule associated with dysmenorrhea, which is increased during dysmenorrhea.
Changes in β-endorphin level | six months
  β-endorphin is a marker molecule associated with dysmenorrhea, which is increased during dysmenorrhea.
Changes in Nitric Oxide level | six months
  NO is a marker molecule associated with dysmenorrhea, which is reduced during dysmenorrhea.
Changes in endothelin level | six months
  Endothelin is a marker molecule associated with dysmenorrhea, which is increased during dysmenorrhea.

CONTACTS AND LOCATIONS:
Overall Officials: Honglan Zhu, M.D, Principal Investigator — Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Proctor M, Farquhar C. Diagnosis and management of dysmenorrhoea. BMJ. 2006 May 13;332(7550):1134-8. doi: 10.1136/bmj.332.7550.1134. No abstract available. PMID 16690671
- [Background] Nasir L, Bope ET. Management of pelvic pain from dysmenorrhea or endometriosis. J Am Board Fam Pract. 2004 Nov-Dec;17 Suppl:S43-7. doi: 10.3122/jabfm.17.suppl_1.s43. PMID 15575029
- [Background] Latthe P, Latthe M, Say L, Gulmezoglu M, Khan KS. WHO systematic review of prevalence of chronic pelvic pain: a neglected reproductive health morbidity. BMC Public Health. 2006 Jul 6;6:177. doi: 10.1186/1471-2458-6-177. PMID 16824213
- [Background] Jamieson DJ, Steege JF. The prevalence of dysmenorrhea, dyspareunia, pelvic pain, and irritable bowel syndrome in primary care practices. Obstet Gynecol. 1996 Jan;87(1):55-8. doi: 10.1016/0029-7844(95)00360-6. PMID 8532266
- [Background] Banikarim C, Chacko MR, Kelder SH. Prevalence and impact of dysmenorrhea on Hispanic female adolescents. Arch Pediatr Adolesc Med. 2000 Dec;154(12):1226-9. doi: 10.1001/archpedi.154.12.1226. PMID 11115307